CLINICAL TRIAL: NCT06643598
Title: Virtual Abecedarian Approach (A2) For IPNH-NDCP (Infants With Perinatal Neurological Histories - At Risk for Neurodevelopmental Disabilities or Cerebral Palsy)
Brief Title: Virtual A2 Study for At Risk Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-1658; Protocol Version 6/26/2025 (Other: UW Madison); A535100 (Other: UW Madison)
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: Hypoxic Ischaemic Encephalopathy (HIE); Premature Birth; Cerebral Palsy; Neurological Disorder
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Premature Birth; Cerebral Palsy; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care Provided (No Intervention): In the No Intervention condition, at-risk children will receive the current standard of care, and no intervention.
- Virtual Abecedarian Approach Intervention (Experimental): In the Virtual Abecedarian Approach Intervention, children will partake in the Abecedarian Approach Intervention through a virtual format.
  Interventions: Behavioral: Abecedarian Approach
- Feasibility Group (Experimental): Participants will be in fewer sessions in order to assess whether the intervention is accepted by the parents.
  Interventions: Behavioral: Abecedarian Approach

INTERVENTIONS:
Behavioral: Abecedarian Approach — The Abecedarian Approach is an early childhood behavioral education program that aims to improve the learning and cognitive development of children in high-risk or at-risk communities. This study will test the efficacy of implementing this approach in a virtual format.
  Arms: Feasibility Group; Virtual Abecedarian Approach Intervention

SUMMARY:
The goal of this behavioral-interventional study is to learn if the Abecedarian Approach implemented virtually for children ages 0-5 with a history of Hypoxic Ischaemic Encephalopathy (HIE) and/or premature birth produces the same effects as when administered at in-person facilities.

ELIGIBILITY:
Inclusion Criteria:

1. IPNH-NDCP patients, including:

   * Term-born children diagnosed during the neonatal period with hypoxic-ischemic encephalopathy, or
   * premature children (born at less than 28 weeks gestational age).
2. Parent or legal guardian will also be enrolled as a participant
3. Parents must be English-speaking (able to provide consent and complete questionnaires).

Exclusion Criteria:

1. Not suitable for study participation due to other reasons at the discretion of the investigator.
2. Infants with chromosomal abnormalities, genetic syndromes (for example, such as Down Syndrome or Trisomy18) and major congenital malformations will be excluded.
3. Infants with vision impairment will also be excluded from the study, as our study procedures do require intact vision to be able to complete.
4. For parents or legal guardians, there are no exclusion criteria.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Parent Satisfaction Questionnaire | Assessed at end of treatment (up to 60 months)
  Questionnaire measuring parent satisfaction with the intervention and effects given at the end of the virtual program. Responses as measured by answering either strongly agree, agree, disagree or strongly disagree. Responses will be measured at the end of the intervention at 60 months and reported as participant counts.
Number of Sessions Attended | Assessed biweekly from enrollment to end of treatment (up to 260 weeks)
  We will be taking attendance of sessions to measure parent compliance with the virtual program. Attendance will be taken for each live session (every other week) for the entire period of enrollment (260 weeks).

SECONDARY OUTCOMES:
Bayley Assessment | Data collected at 12, 24, 36, 48 and 60 month time points
  The Bayley is a cognitive and motor assessment conducted by an interventionalist to assess a child's development in these domains. The highest possible score on a subtest or subdomain is 19, and the lowest score is 1. Scores from 8-12 are considered average.
Behavior Reporting Inventory of Executive Function - Preschool Version (BRIEF-P) | Data collected at the 24, 36, 48 and 60 month time points
  Behavior is reported in the BRIEF-P. Behaviors reported by parents can be used to predict later executive function exhibited by children. List of statements provided about child's behavior, parent will answer whether this is never a problem (N), sometimes a problem (S), and often a problem (O). Responses reported as participant counts, answering N more often is considered a better score.
Pediatric Quality of Life Inventory (PedsQL) | Data collected at 24, 36, 48 and 60 month time points
  The PedsQL is an inventory of statements scored by reverse-scoring responses to a 5-point Likert scale and then transforming them to a 0-100 scale. A higher score indicates a better quality of life.
Early Executive Functions Questionnaire (EEFQ) | Data collected at 12 and 24 month time points
  A questionnaire is given to parents that assesses what executive functions children are exhibiting. More functions exhibited means further along in executive function development. EEFQ consists of 31 tasks parent is scoring child on, there are 7 options they can choose from regarding how that child performs the task, and in turn are scored 1-7 on the task. Tasks listed as designed to measure cognitive executive function, which should be increasing with age, higher scores are indicative of higher cognitive executive function.
NIH Baby/Infant and NIH Pediatric Toolbox | Data collected at 12, 24, 36, 48 and 60-month time points
  A set of tests designed by the NIH administered electronically to children to assess attention, executive function, learning, memory, language, and numeracy/math. A higher early childhood composite score indicates better performance and more of the concept being measured. Early childhood composite score - 100 is the standard, ranges from 70 (extremely low functioning) -130 (extremely high functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Carrasco McCaul, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States